CLINICAL TRIAL: NCT06683911
Title: Comparison of the Postoperative Effects of Opioid-Free Anesthesia and Opioid-Based Anesthesia in Patients Undergoing Open-Heart Surgery With Cardiopulmonary Bypass
Brief Title: Opioids Continue to Play a Primary Role in the Management of Perioperative Pain Due to Opioid-Free Anesthesia in Open Heart Surgery.
Acronym: Opioid-Free
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Seda Kurtbeyoğlu, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: Opioid-Free Anesthesia
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Undergoing Open-Heart Surgery
Keywords: Open-Heart Surgery, opioid free anesthesia
MeSH Terms: interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid free anaesthesia: İnduction = 1 mg/kg lidocaine, 2-3 mg/kg propofol, 15 mg/kg magnesium, 1 mcg/kg dexmedetomidine (over 10 minutes), and a 0.6 mg/kg rocuronium.1 g acetaminophen, 4 mg ondansetron.
  Blocks will include bilateral transverse thoracic muscle plane block and/or bilateral serratus anterior plane block with 0.5% bupivacaine (max 2 mg/kg) under ultrasound guidance.
  Intravenous dexmedetomidine (0.1-1.4 mcg/kg/hr), lidocaine (0.5-1 mg/kg/hr), magnesium (1-10 mg/kg/hr), and propofol (1.5-12 mg/kg/hr) infusions will be adjusted based on hemodynamic parameters to achieve a target BIS value of 40-60.
  if: heart rate <80 and blood pressure >140/90 mmHg, urapidil heart rate >80 and blood pressure >140/90 mmHg, esmolol heart rate <50, atropine mean arterial pressure <60 mmHg, ephedrine will be administered.
  Local infiltration anesthesia will be administered through a catheter placed at the end of surgery, using bupivacaine at a concentration=2mg/ml and dosage=1.5 mg/kg/24 hours
  Interventions: Drug: non Opioids
- opioid anaesthesia: İnduction = 1 mcg/kg remifentanil and/or 1-5 mg fentanyl, 2-3 mg/kg propofol, intravenous 1 mg/kg lidocaine, 2-3 mg/kg propofol, and a 0.6 mg/kg rocuronium.1 g acetaminophen, 4 mg ondansetron.
  Blocks will include bilateral transverse thoracic muscle plane block and/or bilateral serratus anterior plane block with 0.5% bupivacaine (max 2 mg/kg) under ultrasound guidance.
  Intravenous remifentanil (0.02-2 mcg/kg/hr) and propofol (1.5-12 mg/kg/hr) infusions will be adjusted based on hemodynamic parameters to achieve a target BIS value of 40-60.
  if: heart rate <80 and blood pressure >140/90 mmHg, urapidil heart rate >80 and blood pressure >140/90 mmHg, esmolol heart rate <50, atropine mean arterial pressure <60 mmHg, ephedrine will be administered.
  Local infiltration anesthesia will be administered through a catheter placed at the end of surgery, using bupivacaine at a concentration=2mg/ml and dosage=1.5 mg/kg/24 hours
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: non Opioids — It is planned to avoid opioid side effects by applying opioid-free anesthesia during the perioperative period.
  Other Names: opioid anaesthesia
  Groups: opioid free anaesthesia
Drug: Opioid — Routine general anesthesia in cardiac surgery
  Groups: opioid anaesthesia

SUMMARY:
Due to their superior efficacy in analgesia, opioids continue to play a primary role in the control of intraoperative and postoperative pain. Fentanyl, remifentanil, morphine, and tramadol are commonly used opioids during the perioperative period in cardiac surgery. However, the use of opioids requires monitoring, caution, and expertise due to their adverse effects, such as myocardial depression, prolonged respiratory depression, constipation, nausea and vomiting, itching, and dependence. To avoid the side effects caused by opioids, new opioid-free anesthesia protocols have been developed. In addition to avoiding unwanted opioid-related side effects, opioid-free anesthesia provides other benefits, such as rapid postoperative recovery, improvement in postoperative pain scores, enhancement in inflammation parameters, and reduction in postoperative delirium. In opioid-free anesthesia protocols, medications such as dexmedetomidine, magnesium sulfate, lidocaine, ketamine, gabapentin (preoperative and postoperative), dexamethasone, acetaminophen, esmolol, and urapidil are used alongside regional anesthesia techniques to control pain and sympathetic activity.

In this study, patients undergoing elective cardiopulmonary bypass surgery will be included. Procedures will be conducted according to our clinic's routine protocol with monitored general anesthesia induction. Patients included in the study will receive regional blocks and local infiltration anesthesia, which are routine in our clinic. The anesthesia teams, working with the same surgical team in our clinic, will administer either opioid-free anesthesia or anesthesia with opioids. During the perioperative period, the clinicians involved in the study will only observe the patients and record data without intervening in the anesthesia practices.

In this study, our primary aim is to compare the effects of opioid anesthesia and opioid-free anesthesia on postoperative recovery in patients who are provided with multimodal analgesic control through fascial plane blocks and continuous local infiltration anesthesia during the perioperative period. Our secondary objectives are to investigate the effects of opioid-free anesthesia on intensive care and hospital stays, postoperative delirium, inflammation parameters, postoperative surgical complications, arrhythmia, total drug doses used, cost, and patient satisfaction.

DETAILED DESCRIPTION:
Due to their superior efficacy in analgesia, opioids continue to play a primary role in the control of intraoperative and postoperative pain. Fentanyl, remifentanil, morphine, and tramadol are commonly used opioids during the perioperative period in cardiac surgery. However, the use of opioids requires monitoring, caution, and expertise due to their adverse effects, such as myocardial depression, prolonged respiratory depression, constipation, nausea and vomiting, itching, and dependence. To avoid the side effects caused by opioids, new opioid-free anesthesia protocols have been developed. In addition to avoiding unwanted opioid-related side effects, opioid-free anesthesia provides other benefits, such as rapid postoperative recovery, improvement in postoperative pain scores, enhancement in inflammation parameters, and reduction in postoperative delirium. In opioid-free anesthesia protocols, medications such as dexmedetomidine, magnesium sulfate, lidocaine, ketamine, gabapentin (preoperative and postoperative), dexamethasone, acetaminophen, esmolol, and urapidil are used alongside regional anesthesia techniques to control pain and sympathetic activity.

In this study, patients undergoing elective cardiopulmonary bypass surgery will be included. Procedures will be conducted according to our clinic's routine protocol with monitored general anesthesia induction. Patients included in the study will receive regional blocks and local infiltration anesthesia, which are routine in our clinic. The anesthesia teams, working with the same surgical team in our clinic, will administer either opioid-free anesthesia or anesthesia with opioids. During the perioperative period, the clinicians involved in the study will only observe the patients and record data without intervening in the anesthesia practices.

In this study, our primary aim is to compare the effects of opioid anesthesia and opioid-free anesthesia on postoperative recovery in patients who are provided with multimodal analgesic control through fascial plane blocks and continuous local infiltration anesthesia during the perioperative period. Our secondary objectives are to investigate the effects of opioid-free anesthesia on intensive care and hospital stays, postoperative delirium, inflammation parameters, postoperative surgical complications, arrhythmia, total drug doses used, cost, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80
* ASA 1, 2, or 3 status
* Will undergo open-heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* Under 18 years of age
* Over 80 years of age
* Patients with signs of severe organ failure (e.g., kidney or liver failure)
* ASA classification of 4 or higher
* BMI > 40
* Left ventricular ejection fraction < 25%
* Patients with severe arrhythmia
* Patients with severe valve disease
* Aortic surgery
* Preoperative intubation
* Preoperative life support dependency
* Limited preoperative cooperation
* Failed block attempts
* Allergy to any drugs used in the study
* Patients with severe neurological dysfunction
* Patients with contraindications for blocks

Patients who were intubated for more than 12 hours were excluded from the study. Patients who required IABP or ECMO during the perioperative period were excluded from the study. Patients with postoperative cerebrovascular disease and those requiring sedation in the postoperative period were also excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 with ASA 1, 2, or 3 status who undergo open-heart surgery with cardiopulmonary bypass and consent to participate in the study by signing the informed consent form.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
extubation time | postoperative 7 days
  During routine patient visits, the patient's extubation time will be recorded.
mobilization | postoperative 7 days
  During routine patient visits, the patient's first mobilization time will be recorded.
first bowel movement | postoperative 7 days
  During routine patient visits, the patient's first bowel movement in the postoperative period will be recorded and documented.
vomiting | postoperative 1 days
  The patient is questioned and recorded to determine the frequency of opioid side effects during hospital visits.The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and vomiting will be assessed. If the patient has vomited, the number of times they have vomited will be asked and recorded. The total number of times the patient has vomited within 24 hours will be documented.
nausea | postoperative 1 days
  The patient is questioned and recorded to determine the frequency of opioid side effects during hospital visits. The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and their nausea will be assessed. The patient will be asked to provide a number from 0 to 10 to rate the severity of their nausea, and the response will be recorded. 0 means no nausea, and 10 means severe nausea.
Itching | postoperative 1 days
  The patient is questioned and recorded to determine the frequency of opioid side effects during hospital visits. The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and itching will be assessed.
visual analog scale | postoperative 7 days
  The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and their pain will be assessed. The patient will be asked to provide a number from 0 to 10 to rate the intensity of their pain, and the response will be recorded. 0 means no pain, and 10 means unbearable severe pain.
opening eyes first time | postoperative 1 days
  The time when the patient first opens their eyes during the ward round is noted and recorded.
Shivering | postoperative 1 days
  The patient is questioned and recorded to determine the frequency of opioid side effects during hospital visits. The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and shivering will be assessed.
additional analgesics | postoperative 1 days
  It will be assessed whether there is a need for additional analgesics within the first 24 hours. If additional analgesics are required, it will be recorded whether NSAIDs (Non-Steroidal Anti-Inflammatory Drugs) were administered. If they were, the number of times the required and dosage of drug they were given will be noted. It will be recorded whether tramadol was administered. If it was, the number of times it was given and the required dosage in milligrams (mg) will be noted.
The Behavioral Pain Scale (BPS) | postoperative 1 days
  Intubated patients will be assessed at 0,3,6,12,24 hours; using the following criteria, and the total score will be recorded
  Facial expression Relaxed=1 Partially tightened (e.g., brow lowering)=2 Fully tightened (e.g., eyelid closing)=3 Grimacing=4
  Upper limb movements No movement=1 Partially bent=2 Fully bent with finger flexion=3 Permanently retracted=4
  Compliance with mechanical ventilation Tolerating movement=1 Coughing but tolerating ventilation for most of the time=2 Fighting ventilator=3 Unable to control ventilation=4

SECONDARY OUTCOMES:
glascow coma scale | postoperative 7 days
  0,3,6,12 and 24.hour glascow coma scale will be recorded.
  1. Eye Opening (E):
     * 4: Spontaneous
     * 3: To speech
     * 2: To pain
     * 1: No response
  2. Verbal Response (V):
     * 5: Oriented
     * 4: Confused conversation
     * 3: Inappropriate words
     * 2: Incomprehensible sounds
     * 1: No response
  3. Motor Response (M):
     * 6: Obeys commands
     * 5: Localizes pain
     * 4: Withdrawal
     * 3: Flexion to pain (decorticate posture)
     * 2: Extension to pain (decerebrate posture)
     * 1: No response
  Total Score:
  * The scores from each of the three categories are added together.
critical care length of stay | postoperative 7 days
  critical care length of stay will be recorded.
hospital length of stay | postoperative 7 days
  The hospital length of stay will be recorded.
QOR-15 | postoperative 7 days
  The QOR-15 index was used to assess patient satisfaction. A questionnaire containing 15 questions related to patient recovery is administered to patients 24 hours after extubation. For each question, patients are asked to rate their answers on a scale from 0 to 10. The total score is recorded.
  0 = Never 10 = Always

CONTACTS AND LOCATIONS:
Overall Officials: Seda Kurtbeyoglu, doctor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mulier JP. Is opioid-free general anesthesia for breast and gynecological surgery a viable option? Curr Opin Anaesthesiol. 2019 Jun;32(3):257-262. doi: 10.1097/ACO.0000000000000716. PMID 31045633
- [Result] Chanowski EJP, Horn JL, Boyd JH, Tsui BCH, Brodt JL. Opioid-Free Ultra-Fast-Track On-Pump Coronary Artery Bypass Grafting Using Erector Spinae Plane Catheters. J Cardiothorac Vasc Anesth. 2019 Jul;33(7):1988-1990. doi: 10.1053/j.jvca.2018.10.012. Epub 2018 Oct 13. No abstract available. PMID 30424939